CLINICAL TRIAL: NCT04815577
Title: Evolution of Cardiopulmonary Fitness in Children With Congenital Heart Disease : a Longitudinal Multi-center Study
Brief Title: Evolution of Cardiopulmonary Fitness in Children With Congenital Heart Disease
Acronym: Follow-Heart
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0476
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Congenital Heart Disease
Keywords: Congenital heart disease; VO2max; Cardio-pulmonary exercise test
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CHD group: The CHD group is made up of the children included in the first study. From these 496 children with CHD, children with a second CPET more than one year from the first referral CPET were included. If several CPETs were performed in the follow-up, we retain the most distant CPET from the first, excluding the CPETs that were performed after a cardiopulmonary rehabilitation program implemented in the region in 2018. The group corresponding to the first CPET was called. Among the initial 496 children, if patients had not had a second CPET, the cause was indicated. As a reminder, the patients included in the initial study were aged 5-18 years old and they were referred by their paediatric cardiologists to one of the two CPET laboratories after their annual medical check-up. The anatomical and clinical classification of congenital heart diseases was used to define the type of malformation. The demographic, clinical, echocardiographic data were collected during the first CPET.
- Controle: The controle Group consisted of children referred for nonsevere functional symptom linked to exercise (murmur, palpitations or dyspnea) or for a medical sports certificate. We included controlled children from 2015 to 2020 period who will be added to the controlled patients of the initial study. These patients only had one CPET.

SUMMARY:
With an incidence of 0.8 %, congenital heart disease (CHD) is the leading cause of congenital anomalies at birth. Medical advances in CHD have transferred the mortality from childhood to adulthood and today there are more adults with CHD than children. After focusing on survival, more attention is being given to health-related quality of life and secondary prevention in this population where warning signals are launched on the risk of sedentary lifestyle, obesity, cardiovascular risk 1.

The cardiopulmonary exercise test (CPET), which is a non-invasive and dynamic examination, is becoming the gold standard to the follow-up 2 of these patients by allowing to quantify disease severity, to evaluate the quality of life 3, to give important prognostic information on functional capacity and haemodynamic response 4, to facilitate a safe decision-making when prescribing exercise programmes and sport participation for these children with CHD 5.

In this context, in a cross-sectional study from 2010 to 2015, the investigators evaluated the cardiopulmonary fitness of children with CHD by comparing them with healthy children 6. In this study, 496 children with CHD compared to 302 healthy children were included. It showed that maximum oxygen uptake (VO2max) and ventilatory anaerobic threshold (VAT) are decreased in CHD children compared to healthy children, clinical determinants of decreased VO2max have been defined for CHD children. This study was proposed, despite the cross-sectional nature, an average decrease in annual VO2max (0,84 ml/kg/min per year) to make pediatric and congenital cardiologist aware of the need to a regular follow up for these patients.

In this new study, the main objective was to know the real evolution of VO2max in these patients from this same cohort, with a longitudinal design, by collecting a new CPET carried out between 2015 and 2020 and compared these results to healthy pediatric population.

The secondary objectives were: to know the evolution of the VAT, to define the clinical determinants in relation to the annual decrease of the VO2max. And to describe the population lost to follow-up in this retrospective study which represents current practice.

DETAILED DESCRIPTION:
Longitudinal multi-center study from November 2010 to September 2020 in two pediatric CPET laboratories (center 1: M3C Regional Pediatric and Congenital Cardiology Centre, Montpellier University Hospital, France; center 2: Pediatric Cardiology and Rehabilitation Centre, Institut-Saint-Pierre, Palavas-Les-Flots, France).

Two groups will be identify: CHD group and control group. The CHD group is made up of the children included in the first study6. From these 496 children with CHD, children with a second CPET more than one year from the first referral CPET were included. If several CPETs were performed in the follow-up, we retain the most distant CPET from the first. The patients included in the initial study were aged 5-18 years old and they were referred by their paediatric cardiologists to one of the two CPET laboratories after their annual medical check-up.

The control group consisted of children referred for a nonsevere functional symptom linked to exercise (murmur, palpitation or dyspnoea) or for a medical sports certificate. These children were classified in the control group only after a completely normal check-up, including physical examination, ECG, echocardiography and spirometry. Children with any chronic disease, medical condition (cardiac, neurological, respiratory, muscular or renal), or medical treatment and those requiring any further specialised medical consultation were not eligible. We included controlled children from 2015-2020 period who will be added to the controlled patients of the initial study6. These patients only had one CPET.

The main objective was to describe the annual evolution in VO2max for patients with CHD compared to control children.

Secondary obectives were :

* describe the annual evolution of ventilatory anaerobic threshold (VAT) for patients with CHD compared to control children.
* define the clinical determinants in relation to the annual decrease of the VO2 max.
* describe the population lost to follow-up in this retrospective study which represents current practice

ELIGIBILITY:
Inclusion criteria for CHD group :

- children with CHD included in the first study carried out from 2010 to 2015 6 and who have had at least 1 CPET 1 year after the first.

Inclusion criteria for control group :

* children referred for a nonsevere functional symptom linked to exercise (murmur, palpitation or dyspnoea) or for a medical sports certificate.
* completely normal check-up, including physical examination, ECG, echocardiography and spirometry.

Exclusion criteria for control group:

* Children with any chronic disease, medical condition (cardiac, neurological, respiratory, muscular or renal)
* Children with any medical treatment
* Children requiring any further specialised medical consultation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * Children with congenital heart disease with 2 CPET separated at least by 1 year
  * Controlled children with completely normal check-up, including physical examination, ECG, echocardiography and spirometry
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
to give the annual evolution in VO2max for patients with CHD compared to control children | more than 1 year (maximum 8 years)
  comparison of the VO2max value in ml/kg/min between point 1 and point 2 (greater than 1 year) and report the value per year. These results will be compared to evolution of VO2max in controlled children.

SECONDARY OUTCOMES:
to give the annual evolution in VAT for patients with CHD compared to control children | more than 1 year (maximum 8 years)
  comparison of the VAT value in ml/kg/min between point 1 and point 2 (greater than 1 year) and report the value per year. These results will be compared to evolution of VO2max in controlled children.
correlation between clinical determinants and annual decrease of the VO2 max in the CHD group | more than 1 year (maximum 8 years)
  with multivariate analysis, we will look for the correlation between the clinical determinants (collected during the first CPET) and the annual decreased of VO2max in CHD group.
description of the population lost to follow-up in this retrospective study which represents current practice | more than 1 year (maximum 8 years)
  description of demographic data and severity of CHD

CONTACTS AND LOCATIONS:
Overall Officials: Arthur GAVOTTO, MD, Principal Investigator — University Hospital, Montpellier; Pascal AMEDRO, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Background] Amedro P, Mura T, Matecki S, Guillaumont S, Requirand A, Jeandel C, Kollen L, Gavotto A. Use of new paediatric VO2max reference equations to evaluate aerobic fitness in overweight or obese children with congenital heart disease. Eur J Prev Cardiol. 2023 Nov 30;30(17):1865-1873. doi: 10.1093/eurjpc/zwad201. PMID 37314435
- [Derived] Gavotto A, Ladeveze M, Avesani M, Huguet H, Guillaumont S, Picot MC, Requirand A, Matecki S, Amedro P. Aerobic fitness change with time in children with congenital heart disease: A retrospective controlled cohort study. Int J Cardiol. 2023 Jan 15;371:140-146. doi: 10.1016/j.ijcard.2022.09.068. Epub 2022 Sep 29. PMID 36181952